CLINICAL TRIAL: NCT05554276
Title: Neoadjuvant Chemotherapy Combined With PD-1 Antibody + Radical Radiotherapy in Unresectable Locally Advanced Cervical Cancer Patients
Brief Title: Neoadjuvant Chemotherapy Combined With PD-1 + Radical Radiotherapy in Locally Advanced Cervical Cancer
Acronym: PD-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojing Yang, Principal Investigator, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSH06R101
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Neoadjuvant Chemotherapy; PD-1 Antibody; Radiotherapy; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neoadjuvant chemotherapy+ PD-1 antibody + radical radiotherapy (Experimental): All patients received three cycles of 21 days each, with chemotherapy on day 1 (nab-paclitaxel 150 mg/m2 plus cisplatin 75 mg/m2) and camrelizumab 200 mg, followed by radical radiotherapy.
  Interventions: Combination Product: neoadjuvant chemotherapy combined with PD-1 antibody + radical radiotherapy

INTERVENTIONS:
Combination Product: neoadjuvant chemotherapy combined with PD-1 antibody + radical radiotherapy — All patients received three cycles of 21 days each, with chemotherapy on day 1 (nab-paclitaxel 150 mg/m2 plus cisplatin 75 mg/m2) and camrelizumab 200 mg, followed by radical radiotherapy.

SUMMARY:
Based on various external factors and differences in the basic characteristics of patients, in my country, it is not clear whether concurrent chemoradiotherapy can achieve optimal therapeutic effect in patients with pathologically diagnosed stage IIB or above locally advanced cervical cancer. Under the limitations of radiotherapy and surgery conditions in the region, some patients will try neoadjuvant chemotherapy combined with PD-1 antibody therapy before standard radiotherapy, hoping to reduce cancer focus and reduce infiltration. Thereby reducing the scope of radiotherapy, better ensure the efficacy of late radiotherapy and chemotherapy and reduce the side effects of radiotherapy. Judging from the review of such patients, neoadjuvant chemotherapy combined with PD-1 antibody therapy + radical radiotherapy seems to have certain efficacy and tolerance in the near future as expected. No statistical analysis has been done on the long-term survival of patients. This topic intends to treat inoperable locally advanced cervical cancer patients with neoadjuvant chemotherapy combined with PD-1 antibody + radical radiotherapy, and explore the treatment-related toxic and side effects and efficacy of neoadjuvant chemotherapy combined with PD-1 antibody + radical radiotherapy. It is hoped that through this study, it will provide a reference for the comprehensive treatment of inoperable locally advanced cervical cancer that has been pathologically diagnosed in the future.

DETAILED DESCRIPTION:
3.1 Overall study design and planning This study is a prospective, single-arm, phase II, single-center study. Eligible patients with locally advanced cervical cancer entered the trial arm, and all patients received three cycles of 21 days each, with chemotherapy on day 1 (nab-paclitaxel 150 mg/m2 plus cisplatin 75 mg/m2) and camrelizumab 200 mg, followed by radical radiotherapy. Treatment-related acute events were recorded during treatment. Survival period was followed up after the end of treatment, so far the trial treatment ended. (See the following test flow diagram for details).

Schematic diagram of the test process:

3.2 Study population 3.2.1 Selection criteria

1. Age 18-70 years old;
2. Histologically diagnosed as cervical squamous cell carcinoma; clinical evaluation cannot be surgically removed;
3. According to the 2018 International Federation of Obstetrics and Gynecology (FIGO) cervical cancer staging for locally advanced patients, including inoperable stage IIB, IIIA, IIIB, IIIC, IVa;
4. No previous treatment for cervical cancer;
5. According to RECIST version 1.1 criteria, there is at least one evaluable target lesion;
6. ECOG fitness status is 0-1 points;
7. The function of major organs is normal, that is, the following criteria are met:

<!-- -->

1. The standard of blood routine examination must meet: (no blood transfusion within 14 days)

   1. Hb≥90g/L:
   2. ANC≥1.5x10^9/L;
   3. PLT≥80x10^9/L;
2. The biochemical examination shall meet the following standards

   1. BIL < 1.25 times the upper limit of normal (ULN);
   2. ALT and AST < 2.5xULN;
   3. Serum Cr≤ULN, endogenous creatinine clearance rate>50ml/min (Cockcroft-Gaut formula); 8. Sign written informed consent before any trial-related activities; 9. The researcher judges that the research protocol can be followed; 10. Patients who are willing and able to comply with visiting arrangements, treatment plans, laboratory tests and other research procedures.

3.2.2 Exclusion criteria

1. Previously received anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibodies (including ipilimumab) or specifically targeted to T cell costimulation or immune checkpoints Immunotherapy of any other antibody or drug of the pathway; 2. Major surgery ≤4 weeks before enrollment; 3. Those who have been confirmed to be allergic to PD-1 antibody or its excipients; 4. Any active autoimmune disease or history of autoimmune disease (eg, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (hormone replacement therapy is effective) can be included later), etc.: patients with vitiligo or asthma who have been completely relieved in childhood, do not require any intervention in adulthood, and require medical intervention with bronchodilators can be included); 5. Previous or concomitant other malignancies (except those that have been cured, cancer-free survival for more than 5 years, such as skin basal cell carcinoma and papillary thyroid carcinoma, etc.); 6. Uncontrolled cardiac clinical symptoms or diseases, such as: (1) NYHA II or higher heart failure (2) unstable striatal pain (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular Patients with arrhythmia requiring clinical intervention; 7. Subjects requiring systemic treatment with corticosteroids (>10mg/day prednisone efficacy dose) or other immunosuppressive agents within 14 days prior to administration of study drug, inhalation or topical are allowed in the absence of active autoimmune disease Adrenal hormone replacement with steroids and doses >10 mg/day of prednisone at therapeutic doses; 8. Active infection requiring treatment; 9. Suffering from congenital or acquired immunodeficiency (such as HIV infection), active hepatitis B (HBV-DNA≥104 (copy number/ml or 2000IU/ml) or hepatitis C (positive for hepatitis C antibody, and HCV-RNA higher than the analytical method) detection limit); 10. The patient has received other treatments prior to the patient's visit; 11. Received live vaccine within 4 weeks prior to initiation of study treatment; 12. Known history of psychotropic substance abuse, alcohol or drug abuse; 13. pregnant or breastfeeding women; 14. According to the investigator's judgment, the subjects have other factors that may cause them to be forced to terminate the study halfway, such as suffering from other serious diseases (including mental diseases) that require concomitant treatment, severely abnormal laboratory test values, and family or social factors. to the safety of subjects or the collection of trial data; 15. Active pulmonary tuberculosis; 16. Serious infection (including but not limited to hospitalization due to complications of infection, bacteremia or severe pneumonia) occurred within 4 weeks before the start of study treatment; 17. Received systemic immunostimulatory drug treatment (including but not limited to interferon or interleukin-2) within 4 weeks before starting study treatment or within 5 drug half-lives (select the longer of the two).

3.3 The number of cases and the method of grouping This study is a single-arm study, null hypothesis: π≤δ. Alternative hypothesis: π>δ (π is the curative effect index rate of the experimental group). The sample size was calculated based on the exact one-sided binomial test. Assuming that α=0.05, 1-β=80%, and δ=50%, the curative effect of patients with advanced cervical cancer in the past is about 30%, and the dropout rate is 5%. The required sample size is calculated. Sample size calculations were performed using PASS 15.0.1. A total of 36 patients are planned to be enrolled.

3.4 Experimental drugs All patients received three cycles of chemotherapy and immunotherapy, each of 21 days, of which day 1 received chemotherapy (nab-paclitaxel 150 mg/m2 plus cisplatin 75 mg/m2) and camrelizumab 200 mg. All patients received routine antiemetic prophylaxis in each cycle, including 12 mg dexamethasone (intravenous) on day 1 and 8 mg on days 2-4. Definitive radiation therapy (including external beam and/or brachytherapy) was administered 1 to 4 weeks after completion of three cycles of neoadjuvant therapy.

3.5 Study procedures and related examinations Screening period: blood, liver and kidney function, cellular immune index, tumor index, HPV status, pelvic MRI, chest CT, abdominal ultrasound, superficial lymph node ultrasound, PD-L1 comprehensive positive score and patient quality of life self-assessment scale SF-36 score.

Selected treatment period: blood, liver and kidney function, and cellular immune indexes 1-3 days before and 1-7 days after each cycle of neoadjuvant chemotherapy and immunotherapy; re-examination after 2 cycles of neoadjuvant therapy, before radiotherapy, and after radiotherapy Local pelvic MRI examination; patient quality of life self-assessment scale SF-36 score every 3 weeks; treatment-related acute events were recorded during treatment.

Follow-up: 1 month, 3 months, 6 months, 1 year, 2 years, 5 years after treatment, blood, liver and kidney function, cellular immune index, tumor index, pelvic MRI, chest CT, abdominal ultrasound, superficial lymph node ultrasound, etc. The treatment effect was evaluated; at the same time, the intestinal condition of the patients was followed up to evaluate the incidence of radiation enteritis and cystitis.

3.6 End Point indicators Primary endpoint: Objective Response Rate (ORR): refers to the proportion of patients whose tumors shrink to a certain amount and maintain for a certain period of time (more than 4 weeks), including CR+PR cases. CR (complete remission): disappearance of all target lesions, PR (partial remission): reduction of the sum of the length and diameter of the baseline lesions by ≥30%. ; Secondary endpoints: Safety (incidence of treatment acute AEs, radiation enteritis, radiation cystitis); 2-year DFS and OS, and 5-year DFS and OS.

3.7 Criteria for discontinuation of clinical research

1. The patient himself or his legal representative requests to withdraw from the trial;
2. When a patient has an adverse reaction of grade 3 or above, and the adverse reaction does not improve within a week after comprehensive symptomatic treatment, the study can be terminated in advance by evaluating the efficacy, and the case will be treated as an effectively completed case for statistical analysis;
3. The patient has disease progression (definition of disease progression event: transformation to accelerated phase/blast blast phase or death from any cause).

3.8 Combination of medication and treatment

The concomitant medications and usage conditions that may be used as needed during the study are as follows:

1. When adverse events caused by the trial drug require treatment, symptomatic treatment drugs can be given;
2. When the treatment causes bone marrow suppression such as white blood cells and platelets, relevant drugs can be given symptomatic treatment;
3. When the treatment causes abnormal liver and kidney function, related drugs can be given symptomatic treatment;
4. When the treatment causes diarrhea and abdominal pain, related drugs can be given symptomatic treatment;
5. When the treatment causes vomiting, antiemetics can be given;
6. When the patient has symptoms for other reasons, symptomatic treatment drugs can be used.

All concomitant medications should be recorded and stated on the CRF form. 3.9 Follow-up and medical interventions after the end of the study Blood, liver and kidney function, cellular immune index, tumor index, pelvic MRI, chest CT, abdominal ultrasound, and superficial lymph node ultrasound were measured at 1 month, 3 months, 6 months, 1 year, 2 years, and 5 years after treatment. Further treatment should be given if recurrence or corresponding symptoms occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were pathologically diagnosed with cervical squamous cell carcinoma and were assessed as unresectable.

Exclusion Criteria:

* Any active or present autoimmune disease (eg, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 4 weeks after all treatments
  refers to the proportion of patients whose tumors shrink to a certain amount and maintain for a certain period of time (4 weeks after all treatments), including CR+PR cases. CR (complete remission): disappearance of all target lesions, PR (partial remission): reduction of the sum of the length and diameter of the baseline lesions by ≥30%

SECONDARY OUTCOMES:
Side effects | during the procedure
  incidence of treatment acute AEs, radiation enteritis, radiation cystitis
DFS | year 1 and year 5
  year 1 and year 5 DFS
OS | year 1 and year 5
  year 1 and year 5 OS

CONTACTS AND LOCATIONS:
Overall Officials: Jie Fu, Dr, Study Chair — Shanghai Sixth People's Hospital, Shanghai Jiao Tong University
Locations (1):
- Vitalbeam, Shanghai, China

IPD SHARING:
Plan to Share IPD: No